CLINICAL TRIAL: NCT02364921
Title: Effectiveness of Double-layer Compression Therapy in the Healing of Chronic Venous Ulcers in Primary Health Care. Randomized Clinical Trial
Brief Title: Effectiveness of Double-layer Compression Therapy in the Healing of Chronic Venous Ulcers in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI13/01975
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Venous Ulcers
Keywords: venous ulcer; wound healing; compression bandages
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two-layer compression bandage (Experimental): Two multilayer compression bandage: Usual clinical practice in venous ulcer in wound care in assessing, cleaning, desinfection, debridement and topical treatment.Measure the ankle circumference and choose the correct kit accordingly (ankle size 18-25cm or 25-32cm). Apply one to seven days
  Interventions: Device: Two multilayer compression bandage
- crepe bandage (Active Comparator): Crepe bandage: Usual clinical practice in venous ulcer in wound care. crepe bandage apply one to seven days
  Interventions: Device: Crepe bandage

INTERVENTIONS:
Device: Two multilayer compression bandage — Usual clinical practice in venous ulcer in wound care in assessing, cleaning, desinfection, debridement and topical treatment.
  Compression therapy: a multilayer compression bandage with two layers, suitable for the treatment of venous leg ulcers and to reduce edema chronic venous be used. Apply one two seven days
  Other Names: K2 Urgo
  Arms: Two-layer compression bandage
Device: Crepe bandage — Crepe bandage: Usual clinical practice in venous ulcer in wound care. crepe bandage apply one to seven days
  Arms: crepe bandage

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a multilayer compression bandage (two layers), compared with the crepe bandage, on healing of venous leg ulcers, in patients attended in nursing Primary Care Health Centres, at 12 weeks follow-up.

DETAILED DESCRIPTION:
This study also compares the effectiveness of the multilayer and the crepe bandage, on healing of venous leg ulcers measured by the Resvech 2.0 scale and evaluates improvement in quality of life, measured by the Charing Cross Venous Ulcer Questionnaire (CCVUQ-e) and analyze the sociodemographic, clinical, and treatment factors associated with complete healing of venous ulcers.

Design: Multicentre, controlled, parallel group, randomized clinical trial, with blind evaluation of the response variable.

Setting: Primary Care Health Centres (Madrid). Subjects: Patients with venous leg ulcers, treated by nurses at the participating centres.

Intervention: Experimental group: multilayer compression bandage (two layers). Control group: crepe bandage.

Sample size: 216 patients (108 in each group) Variables:Main: Complete healing after 12 weeks follow-up. Secondary: Degree of healing (Resvech 2.0). Quality of life (CCVUQ-e). Adverse reactions. Related to the healing process: comorbidities, topical and systematic treatments, exercise, BMI. Prognostic factors: location, number and duration of ulcer. Sociodemographic factors Data analysis: By intention to treat. Comparative analysis of the two groups (chi-squared or t-test). Effectiveness analysis sing Kaplan-Meier, log rank test and cox regression analysis

ELIGIBILITY:
Inclusion Criteria:

* People With a diagnosis of chronic venous ulcer over six weeks duration.
* Presence of a larger Ankle Arm index (ABI) of 0.8 and less than 1.3.
* People Able to follow the trial own demands, able to understand the questionnaires, with no intention of moving and localizable for the duration of the study.
* That give written informed consent to participate

Exclusion Criteria:

* Patients diagnosed with poorly controlled diabetes mellitus (last HbA1c greater than 7).
* In Antineoplastic therapy.
* Decompensated heart -insufficience .
* Dermatitis acute phase, at the time of the study.
* Rheumatoid-arthritis.
* Thrombosis Venosa (DVT) in acute phase.
* Patients with mixed ulcers
* Patients who participate simultaneously in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
degree of scarring achieved measured by Resverch 2.0 | twelve weeks
  degree of scarring achieved measured by the questionnaire Resverch 2.0

SECONDARY OUTCOMES:
Quality of Life measured by Charing Cross Venous Ulcer Questionnaire (CCVUQ-e) | twelve weeks
  Quality of Life measured by the test Charing Cross Venous Ulcer Questionnaire (CCVUQ-e)

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Carmen Folguera, Nurse, Principal Investigator — Gerencia Atención Primaria, Madrid
Locations (1):
- Carmen Folguera, Madrid, Spain

REFERENCES:
- [Derived] Folguera-Alvarez C, Garrido-Elustondo S, Verdu-Soriano J, Garcia-Garcia-Alcala D, Sanchez-Hernandez M, Torres-de Castro OG, Barcelo-Fidalgo ML, Martinez-Gonzalez O, Ardiaca-Burgues L, Solano-Villarrubia C, Lebracon-Cortes PR, Molins-Santos C, Fresno-Flores M, Canovas-Lago MC, Benito-Herranz LF, Garcia-Sanchez MT, Castillo-Pla O, Morcillo-San Juan MS, Ayuso-de la Torre MB, Burgos-Quintana P, Lopez-Torres-Escudero A, Ballesteros-Garcia G, Garcia-Cabeza P, de Francisco-Casado MA, Rico-Blazquez M; ECAMulticapa Group. ECAMulticapa: Effectiveness of double-layered compression therapy for healing venous ulcers in primary care: a Study Protocol. BMC Nurs. 2016 Oct 12;15:58. doi: 10.1186/s12912-016-0179-x. eCollection 2016. PMID 27752238